CLINICAL TRIAL: NCT05057000
Title: Effect of Aerobic Exercises and Nutrition on The Activities of Daily Living and Estrogen Level in Adolescent Girls With Anorexia
Brief Title: Effect of Aerobic Exercises and Nutrition In Adolescent Girls With Anorexia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Badr University (Other)
Responsible Party: Principal Investigator, Mariam Hossam El Ebrashy, Lectruer of physical therapy for women'shealth, Badr University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BUC
Record Dates: First submitted 2021-09-13; First posted 2021-09-27 (Actual); Last update posted 2022-01-04 (Actual); Status verified 2022-01

CONDITIONS: Anorexia in Adolescence
Keywords: anorexia; adolescent girls; areobic exercises
MeSH Terms: conditions — Anorexia | interventions — Exercise; Diet

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): DIET PROGRAM IN ADDITION TO AEROBIC EXRCISES
  Interventions: Other: aerobic exercises + Diet
- Group B (Other): DIET PROGRAM
  Interventions: Other: diet proram

INTERVENTIONS:
Other: aerobic exercises + Diet — Frequency 5-6 days per week Intensity To perform moderate intensity for weight-bearing aerobic exercise Time Goal of 20-30 min per session of moderate-intensity aerobic activity per week
  Arms: Group A
Other: diet proram — diet program for anorexic adolescent girls
  Arms: Group B

SUMMARY:
Randomized control study used to identify the effect of aerobic exercises on the activity of daily living and estradiol serum level in young girls with anorexia

DETAILED DESCRIPTION:
Control group will receive diet program while the study group received the same diet program given to control group in addition to AEROBIC exercise program.

Inclusive criteria

* Thirty girls with anorexia
* BMI ≤ 18 kg/m2
* Age ranged from (14-17 years).
* Exclusive criteria:
* Girls did not receive any exogenous steroid and other treatment which could affect plasma levels of estrogen hormone.
* Exclude any other eating disorders

Data analysis and statistical design:

The collected data will be statistically treated using:

Descriptive statistics.

Inferential statistics using:

Paired t-test.

ELIGIBILITY:
Inclusion Criteria:

* Thirty girls with anorexia
* BMI ≤ 18 kg/m2
* Age ranged from (14-17 years).

Exclusion Criteria:

Girls did not receive any exogenous steroid and other treatment which could affect plasma levels of estrogen hormone.

Ages: 14 Years to 17 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2021-10-05 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2021-12-30 (Estimated)

PRIMARY OUTCOMES:
Estradiol level | 3 months
  blood test

CONTACTS AND LOCATIONS:
Locations (1):
- Badr University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided